CLINICAL TRIAL: NCT05078918
Title: Development and Evaluation of Comprehensive Care Program for Their Return to Normal Life and Community Among Lung Cancer Survivors
Brief Title: Comprehensive Care Program for Their Return to Normal Life Among Lung Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Dong Wook Shin, Professor of Family Medicine, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMC 2021-08-071
Record Dates: First submitted 2021-09-17; First posted 2021-10-15 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer; Lung Neoplasm
Keywords: Lung Cancer; Survivorship; Quality of Life
MeSH Terms: conditions — Lung Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled trial. Control groups will be enrolled first considering contamination of educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive care program (Experimental): Intervention group receiving newly developed comprehensive care program pre- and post-operatively.
  Interventions: Other: Comprehensive care program
- Usual care (Active Comparator): Control group receiving usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Comprehensive care program — Comprehensive care program includes education and re-evaluation process. Education using video-materials to help patients adapt to the new normal before and after surgery. And re-evaluation patient's needs 1 month after surgery and arrangement resources.
  Other Names: Education and re-evaluation process
  Arms: Comprehensive care program
Other: Usual care — Usual care includes encouraging deep breathing and exercise using inspirometer, postoperative early ambulation, giving information at discharge and follow up 1 month after surgery.
  Other Names: Providing usual care
  Arms: Usual care

SUMMARY:
The purpose of this study is to develop a comprehensive care program for their return to normal life and community among lung cancer survivors and evaluate the effectiveness of the program.

DETAILED DESCRIPTION:
Lung cancer patients scheduled for curative surgery will be enrolled in this study. The comprehensive care program will be developed, and provided to the intervention group before and after surgery. Outcomes will be assessed 6 months and 1 year after surgery. To evaluate the effectiveness of the program, a control group will be enrolled first and used as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-small cell lung cancer(NSCLC) and scheduled for curative resection.
* NSCLC with clinical stage Ⅰ-Ⅲ
* Patients who understood the study and gave written informed consent.

Exclusion Criteria:

* Recurred lung cancer
* Patients with extra-pulmonary synchronous double primary cancer.
* Patients with history of other cancer diagnosis or treatment in the last 3 years.

Drop Criteria:

* When surgery was canceled or pathologic stage IV was confirmed after surgery.
* When the tumor was not found to be non-small cell lung cancer, including benign tumor, after surgery
* Withdrawal informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-09-08 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Mental adjustment to cancer at 6 months after surgery | 6 months after surgery
  The Mini-Mental Adjustment to Cancer (Mini-MAC) scale, a short form instrument derived from the MAC and designed to measure coping with cancer. The scale consists of 29 items and 5 sub-dimensions as follows: Fighting spirit, helplessness/hopelessness, anxious preoccupation, fatalism and cognitive avoidance. The mini-MAC is a Likert type scale with four response options: (1) definitely does not apply to me (2) does not apply to me (3) applies to me (4) definitely applies to me.

SECONDARY OUTCOMES:
Quality of life (EORTC QLQ-C30) | Before surgery (baseline) and 1, 6, 12 months after surgery
  The quality of life is assessed by the European Organization for Research Treatment of Cancer Quality of Life Questionnaire core30 (EORTC QLQ-C30). The scale for quality of life is transformed into a score from 0 to 100, derived by 4-point Likert scale. Higher scores represent a better quality of life.
Lung cancer specific symptoms | Before surgery (baseline) and 1, 6, 12 months after surgery
  The symptoms are assessed by the European Organization for Research Treatment of Cancer Quality of Life Questionnaire lung cancer module 13 (EORTC QLQ-LC13). The scale for symptom is transformed into a score from 0 to 100, derived by 4-point Likert scale. Higher scores mean a more burden of disease.
Dyspnea (mMRC) | Before surgery (baseline) and 1, 6, 12 months after surgery
  Dyspnea is measured by the modified Medical Research Council Dyspnea Scale (mMRC). The mMRC scales grade 0 to grade 4, based on the severity of dyspnea.
Dyspnea (CAT) | Before surgery (baseline) and 1, 6, 12 months after surgery
  Dyspnea is also measured by COPD Assessment Test (CAT). Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Unmet Needs | Before surgery (baseline) and 1, 6, 12 months after surgery
  Unmet needs are assessed by the Cancer Survivors' Unmet Needs (CaSUN). There are 5 domains; existential survivorship (14-item), Comprehensive Cancer Care (6-item), Information (3-item), Quality of Life (2-item), Relationships (3-item). It assesses the unmet needs and strength of needs. In this study, only the information domain is investigated.
Anxiety and depression | Before surgery (baseline) and 6, 12 months after surgery
  Anxiety and depression are assessed by the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item instrument that reflects two dimensions; depression (seven items) and anxiety (seven items). Each item is rated on a 4-point scale from 0 to 3, with a maximum of 21 for anxiety and depression.
Physical Activity | Before surgery (baseline) and 1, 6, 12 months after surgery
  Physical activity is assessed by International Physical Activity Questionnaire-7 (IPAQ-7). This questionnaire measures duration (minutes) and frequency (days) of physical activity in the last 7 days.
Mental adjustment to cancer | Before surgery (baseline) and 12 months after surgery
  The Mini-Mental Adjustment to Cancer (Mini-MAC) scale, a short form instrument derived from the MAC and designed to measure coping with cancer. The scale consists of 29 items and 5 sub-dimensions as follows: Fighting spirit, helplessness/hopelessness, anxious preoccupation, fatalism and cognitive avoidance. The mini-MAC is a Likert type scale with four response options: (1) definitely does not apply to me (2) does not apply to me (3) applies to me (4) definitely applies to me.
Distress | Before surgery (baseline) and 1, 6, 12 months after surgery
  NCCN Distress Thermometer & Problem List

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wook Shin, MD., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung W, Ahn A, Lee G, Kong S, Kang D, Lee D, Kim TE, Shim YM, Kim HK, Cho J, Cho J, Shin DW. Supporting Life Adjustment in Patients With Lung Cancer Through a Comprehensive Care Program: Protocol for a Controlled Before-and-After Trial. JMIR Res Protoc. 2024 Feb 13;13:e54707. doi: 10.2196/54707. PMID 38349712